CLINICAL TRIAL: NCT06656533
Title: Improving Insomnia Treatment by Optimizing Timing of RTMS Administration
Brief Title: Optimizing the Timing of RTMS to Enhance the Administration of Insomnia Treatment
Acronym: TREAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrea Goldstein-Piekarski, ASSISTANT PROFESSOR, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76766
Record Dates: First submitted 2024-10-11; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Insomnia
Keywords: Sleep; Insomnia; rTMS Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MORNING GROUP (Experimental): Five participants (21 to 45 years old) experiencing clinically meaningful insomnia symptoms will be enrolled and will receive 10 sessions of right dorsolateral prefrontal cortex (DLPFC) rTMS therapy in the morning over two consecutive weeks.
  Interventions: Other: Repeated Transcranial magnetic stimulation (rTMS)
- EVENING GROUP (Experimental): Five participants (21 to 45 years old) experiencing clinically meaningful insomnia symptoms will be enrolled and will receive 10 sessions of right dorsolateral prefrontal cortex (DLPFC) rTMS therapy in the evening over two consecutive weeks.
  Interventions: Other: Repeated Transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Other: Repeated Transcranial magnetic stimulation (rTMS) — Transcranial Magnetic Stimulation (TMS) involves a procedure where parts of the participants brain will be non-invasively (i.e. indirectly) stimulated by magnetic pulses. These magnetic pulses induce very brief activity in brain areas underlying the TMS coil. TMS will be performed by giving repetitive pulses (rTMS). rTMS has shown promise to reduce cortical hyperexcitability and to improve subjective measures of sleep quality and insomnia symptoms in patients with insomnia disorder. The goal of this study is to optimize the impact of rTMS therapy on sleep outcomes for patients with insomnia disorder.

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has shown to be a promising technique for improving insomnia symptoms and sleep quality. However, the impact of circadian rhythmicity on rTMS sessions and its potential influence on insomnia therapy remains unclear. Moreover, the effect of rTMS on objective sleep parameters is not fully established. The objective of this pilot study is to establish key feasibility and preliminary data that would be used for an R-level grant application focused on optimizing rTMS therapy for insomnia. The investigators will acquire feasibility data from ten adults with Insomnia disorder. Participants will receive ten sessions rTMS over two weeks, either in the morning or evening. Sleep parameters will be assessed before, during, and after completion of rTMS and brain cortical excitability will be collected before rTMS treatment. The investigators aim to 1) evaluate the impact of circadian timing of rTMS sessions on subjective and objective sleep outcomes, 2) assess the time course of improvements in sleep outcomes, and 3) examine the association between sleep outcomes and cortical excitability. The overarching goal of this work is to optimize rTMS therapy for insomnia by investigating the impact of circadian timing on rTMS sessions and assessing potential variations in subjective and objective measures of sleep.

DETAILED DESCRIPTION:
Low frequency (1 Hz) rTMS has shown promise to reduce cortical hyperexcitability and to improve subjective measures of sleep quality and insomnia symptoms in patients with insomnia disorder (ID) (Nardone et al. 2020). However, the few studies to date that have examined the objective measures of sleep parameters using Polysomnography (PSG), have yielded heterogeneous results. The variability in the PSG measures of sleep may potentially be attributed to the effectiveness of rTMS therapy delivered at different times of day because of changes in cortical excitability related across the 24-hour period (Ly et al. 2016) as well as the temporal proximity of the stimulation to sleep. However, the impact of the timing of rTMS administration on improving insomnia has not yet been examined. In this pilot study, the investigators aim to demonstrate the feasibility of the data acquisition using the proposed protocol and to establish preliminary data that would be used in a future R-level grant. Building on this preliminary data, the future R-level grant would be focused on optimizing rTMS therapy for insomnia and sleep quality by manipulating the time of day that the rTMS sessions are delivered. In the following, the investigators will provide their aims for this pilot study.

The investigators' objectives are 1. To assess the impact of morning versus evening administration of rTMS on a) subjective and b) objective sleep outcomes. Here the investigators propose to enroll 10 participants and randomize each to either receive 10 sessions of rTMS over two weeks in the morning or in the evening. This pilot study would provide preliminary time-of-day effects on subjective (sleep diary parameters and insomnia severity) and objective sleep (wristwatch actigraphy and PSG) measures. It characterizes the time course of improvement across the two-week treatment period for a) subjective and b) objective sleep measures. Throughout the multi-week intervention, the investigators will collect subjective and objective sleep measures to characterize the improvement across the two-week period.

Finally, this pilot study would determine whether cortical excitability predicts treatment outcomes. Participants will undergo a TMS-EEG session before rTMS therapy. Cortical excitability will be assessed by measuring TMS-evoked EEG potentials (TEP).

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any racial or ethnic group, aged 25-45 (inclusive)
* Insomnia diagnosis via the DUKE
* Fluent and literate in English
* Written, informed consent
* Reside within 60 miles of Stanford University

Exclusion Criteria:

* Presence of other sleep or circadian rhythm disorders that significantly contribute to their sleep disturbance. The presence of these disorders will be assessed by the DUKE structured interview for sleep disorders.
* No regular use of benzodiazepine, opiate, thyroid, anticonvulsant or antipsychotic medications
* Use of psychotropic medications that would significantly impact sleep, alertness, and no illicit drugs.
* Excessive alcohol consumption (>14 drinks per week or > 4 drinks per occasion)
* Presence of suicidal ideations representing elevated risk as determined by the Beck Depression Inventory (score of > 0 on BDI question #9).
* History of neurological or cardiovascular disorders, brain surgery, electroconvulsive or radiation treatment, brain hemorrhage or tumor, stroke, seizures or epilepsy, diabetes, hypo- or hyperthyroidism, head trauma with loss of consciousness greater than thirty minutes.
* Substance abuse or dependence
* History of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities OR traumatic brain injury in the past two months
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to complete the assessments, or are unable and/or unlikely to follow the study protocols
* Pregnant or breast feeding
* Current or lifetime history of bipolar disorder, PTSD or psychosis or current depression
* Received cognitive behavioral therapy for insomnia within the past year
* Current exposure to trauma, or exposure to trauma within the past 3 months
* Working a rotating shift that overlaps with 2400h
* Individuals who were high risk for sleep apnea on the Berlin Questionnaire and are not CPAP adherent
* Participants with a current psychiatric disorder who are also on medications that significantly increase the risk of seizure. The antidepressants clomipramine, bupropion, maprotiline will be excluded because they are known to increase risk of up to 0.5-2.2% from a population reference range of 0.07- 0.08% in the general population and 0.1-4% in the population of people taking antidepressants.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Insomnia severity index will be collected within one week before and within one week after the 10 sessions (over two weeks) of rTMS therapy.
  Improvement in insomnia symptoms will be assessed using the Insomnia Severity Index (ISI). ISI is a 7-item self-report questionnaire designed to assess the severity of insomnia symptoms and their impact on daily functioning. Each question is scored on a 5-point Likert scale, with ratings from 0 (no problem) to 4 (very severe problem).
Pittsburgh Sleep Quality Index | Pittsburgh Sleep Quality Index will be collected within one week before and within one week after the 10 sessions (over two weeks) of rTMS therapy.
  Improvement in subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). PSQI is a widely used questionnaire that assesses sleep quality and disturbances over one month. It includes seven components and ranges from 0 to 21, with higher scores indicating poorer sleep quality. A score above 5 is generally considered indicative of poor sleep quality.

SECONDARY OUTCOMES:
OBJECTIVE SLEEP MEASURES | EEG sleep parameters will be collected within one week before and within one week after 10 sessions (over two weeks)of rTMS therapy. Actiwatch sleep measures will be collected from one week before the baseline session to the end of the treatment session.
  Changes in sleep parameters, objectively measured using an Electroencephalogram (EEG) and Actiwatch, will be assessed following rTMS therapy. Sleep Efficiency (the percentage of time a person spends asleep compared to the total amount of time they spend in bed), Wake After Sleep Onset (the amount of time a person is awake after falling asleep but before waking up for the day), and Sleep Latency ( the amount of time it takes to fall asleep after turning off the lights) will be calculated from EEG and Actiwatches. Additionally, sleep architecture including time spent in sleep stages and spectral measures will be collected using EEG.
Cortical Excitability | Cortical excitability will be measured during the first therapy session, before the first rTMS therapy.
  Cortical excitability, defined as the strength of cortical neural responses to stimulations, will be assessed by measuring TMS-evoked EEG potentials (TEP).
  Specifically, the amplitude of the change in EEG data after a single TMS pulse in the supplementary motor area will be quantified and associated with changes in sleep measures and insomnia severity index.

CONTACTS AND LOCATIONS:
Locations (1):
- 1070 Arastradero Road, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ly JQM, Gaggioni G, Chellappa SL, Papachilleos S, Brzozowski A, Borsu C, Rosanova M, Sarasso S, Middleton B, Luxen A, Archer SN, Phillips C, Dijk DJ, Maquet P, Massimini M, Vandewalle G. Circadian regulation of human cortical excitability. Nat Commun. 2016 Jun 24;7:11828. doi: 10.1038/ncomms11828. PMID 27339884
- [Background] Nardone R, Sebastianelli L, Versace V, Brigo F, Golaszewski S, Pucks-Faes E, Saltuari L, Trinka E. Effects of repetitive transcranial magnetic stimulation in subjects with sleep disorders. Sleep Med. 2020 Jul;71:113-121. doi: 10.1016/j.sleep.2020.01.028. Epub 2020 Feb 19. PMID 32173186